CLINICAL TRIAL: NCT06043063
Title: Post-procedural Pain Associated With Periurethral Block at Time of Bulkamid Injection for SUI: a Randomized Controlled Trial
Brief Title: Local Anesthesia Before Bulkamid Injection
Acronym: LAB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated prematurely due to meeting safety endpoint defined as 3 participants in the experimental arm requiring termination of in-office procedure due to pain.
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006172
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence; Intrinsic Sphincter Deficiency
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lidocaine; Lidocaine, Prilocaine Drug Combination; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical anesthesia alone (Experimental): 2.5% EMLA cream + intraurethral 2% lidocaine gel for 15 min
  Interventions: Procedure: Topical lidocaine; Procedure: EMLA cream
- Topical anesthesia with periurethral block (Active Comparator): 2.5% EMLA cream + intraurethral 2% lidocaine gel for 15 min
  + periurethral block (5 cc 1% lidocaine or 0.25% bupivacaine at 3 and 9 o'clock to depth of 1.5 cm using 25G needle)
  Block sits for 5 min if lidocaine, 10 min if bupivacaine
  Interventions: Procedure: Topical lidocaine; Procedure: EMLA cream; Procedure: Periurethral block

INTERVENTIONS:
Procedure: Topical lidocaine — Topical anesthetic
  Other Names: Intraurethral 2% lidocaine gel
Procedure: EMLA cream — Topical anesthetic
  Other Names: 2.5%/2.5% EMLA (eutectic mixture of local anesthetics) cream
Procedure: Periurethral block — 5 cc 1% lidocaine or 0.25% bupivacaine at 3 and 9 o'clock (periurethral tissues) to depth of 1.5 cm using 25G needle
  Other Names: 1% lidocaine or 0.25% bupivacaine
  Arms: Topical anesthesia with periurethral block

SUMMARY:
While recommended pre-anesthesia for polyacylamide hydrogel (PAHG, Bulkamid) injections for stress urinary incontinence and intrinsic sphincter deficiency can include intraurethral anesthetic gel with or without periurethral block, there is no existing literature to guide choice of anesthesia. This is a single-blinded randomized control trial to evaluate post-procedure pain with choice of anesthesia before PAHG injection.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old with stress urinary incontinence, intrinsic sphincter deficiency, or stress-predominant mixed urinary incontinence desiring PAHG
* English-speaking
* Scheduled in outpatient clinic or OR without sedation, general, or neuraxial anesthesia

Exclusion Criteria:

* Pregnancy
* Neurogenic bladder
* Pre-existing need for intermittent catheterization or indwelling catheter
* Bladder or urothelial malignancy
* Prior radiation to pelvic floor
* Known allergy/sensitivity to PAHG

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain | Ascertained at end of procedure (withdrawal of cystoscope)
  Visual analog scale for pain uses a scale from 0-10 corresponding to reported pain levels with 0 indicating no pain and 10 indicating most severe pain possible

SECONDARY OUTCOMES:
Duration of procedure | Ascertained at end of procedure (within 5 minutes of withdrawal of cystoscope)
  in seconds
Incomplete bladder emptying | Ascertained on day-of-procedure (within 1 hour of withdrawal of cystoscope)
  Inability to void after procedure
Need for re-injection of PAHG | Assessed at follow-up 2 weeks post-procedure
  Requirement for "top-off" or repeat injection due to persistent symptoms
International Consultation on Incontinence Questionnaire for Urinary Incontinence (ICIQ-UI) | Assessed at baseline and at two-week and twelve-week follow-up visit
  3 items on frequency/quantity of leakage and impact on quality on life (range 0-21 with lower score indicating lower severity of incontinence symptoms and higher score indicating higher severity of incontinence symptoms)
Patient Global Impression of Improvement scale (PGI-I) | Assessed at two-week and twelve-week follow-up visit
  1 item on relative change in symptoms following treatment (range 1-7 with lower score indicating greater improvement in incontinence symptoms following intervention and higher score indicating lower improvement in incontinence following intervention)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Lafayette Medical Centre, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No